CLINICAL TRIAL: NCT01067625
Title: Endoscopic Bariatric Stapling Pilot Study
Acronym: TOGA®
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: Satiety, Inc. (Industry)
Responsible Party: Allan L. Abati, Ph.D., VP, RA/QA and Clinical Programs, Satiety, Inc.
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: TR-0009 Rev F
Record Dates: First submitted 2010-02-10; First posted 2010-02-11 (Estimated); Last update posted 2010-02-11 (Estimated); Status verified 2010-02

CONDITIONS: Obesity
MeSH Terms: conditions — Obesity

ARMS (1):
- TOGA subjects (Experimental)
  Interventions: Device: TOGA® System

INTERVENTIONS:
Device: TOGA® System — Formation of restrictive sleeve via transoral gastric stapling for treatment of obesity

SUMMARY:
This study is a prospective single-arm, multicenter study to evaluate the safety and effectiveness of the TOGA® Procedure for the treatment of morbid obesity.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18 years - 60 years
2. Eligible for bariatric surgery per US National Institute of Health (NIH) guidelines BMI ≥ 40 kg/m2 and < 55 kg/m2, or BMI ≥ 35 kg/m2 with one or more comorbidities. Comorbidities are defined as diabetes, pulmonary disease, cardiac disease, or hypertension [systolic blood pressure of ≥140 mm Hg or diastolic blood pressure ≥ 90 mm Hg (or both) or on treatment for hypertension]
3. History of obesity for at least 2.5 years
4. History of failure with non-surgical weight loss methods.
5. Agree to comply with the substantial dietary restrictions required by the procedure.
6. Understands risks of procedures, agree to follow protocol requirements, including signing informed consent, returning for follow-up visits and completing all required testing, completing diet and behavior modification counseling.

Exclusion Criteria:

1. Patient history of inflammatory disease of the gastrointestinal tract including Crohn's disease or ulcerative colitis.
2. Significant known esophageal disease including grade 3-4 esophagitis, stricture, Barrett's esophagus, esophageal cancer, esophageal diverticulum, nutcracker esophagus, achalasia, esophageal dysmotility.
3. Severe coagulopathy, upper GI bleeding conditions such as esophageal or gastric varices, congenital or acquired telangiectasia.
4. Congenital or acquired anomalies of the GI tract such as atresias or stenoses.
5. Hiatal hernia ≥2cm
6. Severe cardiopulmonary disease or other serious organic disease including HIV or cancer.
7. Currently pregnant or nursing. Potentially childbearing (i.e not post-menopausal or surgically sterilized) and not willing to use an effective method of contraception for the next 12 months.
8. Current alcohol or drug addiction.
9. Mentally retarded or emotionally unstable, or exhibits psychological characteristics which, in the opinion of the investigator or psychologist/psychiatrist, make the subject a poor candidate for this procedure.
10. Previous gastric, esophageal, pancreatic, or bariatric surgery.
11. Infection anywhere in the body at the time of the procedure.
12. Patient history of scleroderma.
13. Thyroid disease which is not controlled with medication.
14. Participating in another ongoing clinical trial in which concomitant diagnosis or therapeutic intervention would adversely affect the integrity of the clinical trial.
15. Known active H-pylori infection.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 200 (Estimated)
Dates: Start 2006-02; Primary Completion 2015-12 (Estimated)

PRIMARY OUTCOMES:
Percent excess weight loss (%EWL) | up to 60 months
Adverse events, including serious adverse events, will be recorded to determine safety | up to 60 months

SECONDARY OUTCOMES:
Improvement in Co-morbidities | up to 60 months
Improvements in other Obesity Measures and Change in Quality Of Life Measures | up to 60 months

CONTACTS AND LOCATIONS:
Locations (2):
- ULB (Universite Libre de Bruxelles) - Erasme Hospital, Brussels, Belgium
- Università Cattolica del Sacro Cuore - Policlinico A. Gemelli, Rome, Italy

REFERENCES:
- [Derived] Familiari P, Costamagna G, Blero D, Le Moine O, Perri V, Boskoski I, Coppens E, Barea M, Iaconelli A, Mingrone G, Moreno C, Deviere J. Transoral gastroplasty for morbid obesity: a multicenter trial with a 1-year outcome. Gastrointest Endosc. 2011 Dec;74(6):1248-58. doi: 10.1016/j.gie.2011.08.046. PMID 22136774